CLINICAL TRIAL: NCT01131598
Title: Acute Lung Injury in Spanish Children
Brief Title: Acute Lung Injury in Children: Epidemiology and Natural History. PEDIATRIC ALIEN.
Acronym: ALIEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Cruces (Other)
Collaborators: Spanish Intensive Care Pediatrician Society (Unknown)
Responsible Party: Jesús Villar and Robert Kacmarek, Spanish Intensive Care Pediatrician Society
Other Study IDs: Acute lung injury in children
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-01

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: ALI; SDRA
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to perform a one-year prospective audit of all Acute lung injury (ALI)and cute respiratory distress syndrome (ARDS) pediatric patients managed in several ICUs in Spain. The investigators intend to collect data from all children (from 1 month to 18 years of age) admitted with or developing ALI/ARDS with the aim to understand the epidemiology and natural history of acute lung injury in the pediatric setting. These ICUs are scattered through the Spain and are representative of the demographic differences across the country.

DETAILED DESCRIPTION:
Acute lung injury (ALI) is a clinical syndrome of rapid onset of non-cardiogenic pulmonary edema manifested clinically by hypoxemia (PaO2/FiO2≤300 mmHg) and bilateral pulmonary infiltrates. When the hypoxemia is severe (PaO2/FiO2≤200 mmHg) it is termed the acute respiratory distress syndrome (ARDS). It represents a significant public health issue. Patients with ALI or ARDS require admission into critical care units for advanced life support and utilize considerable health care resources.

An immense plethora of translational knowledge has been acquired since the first description of ARDS in 1967. At the present, estimates of the incidence of ARDS and ALI in children are unknown. In adults, the estimates of ALI/ARDS incidence have varied widely, and the true magnitude of this health problem still remains unclear. Current estimates of the incidence of adult ALI/ARDS range from 15 to 80 cases per 100.000 population, or almost 40.000 cases per year in Spain. Combined mortality rates for adult ALI/ARDS range between 30-45% but it is not clear whether this figures can be translated in the pediatric population. ALI and ARDS occur as a complication or as the primary cause of critical illness in patients, usually after severe infection or trauma.

Published epidemiological studies on ALI and ARDS in the last 20 years are difficult to compare. Some reports have used different definitions for ALI and ARDS and others have evaluated the incidence during a short period of time (from days to several weeks) and then extrapolated their data to estimates of a one-year incidence. Very few studies have collected information for an entire year, and none of them have evaluated the degree of hypoxemia under standard ventilatory settings, as it has been proposed recently by the HELP Network (Am J Respir Crit Care Med 2007; 176:795-804).

ELIGIBILITY:
Inclusion criteria:

* All patients, age ranging from 1 month to 15 years old
* Must be able to meet the American European Consensus definition of ALI and ARDS(no indication of heart failure or a pulmonary capillary wedge pressure of greater than 18 mmHg, with pulmonary infiltrates in all four quadrants and a PaO2/FIO2 of > 200 to <300 mmHg (ALI) or ? 200 mmHg (ARDS).

Exclusion criteria:

* Younger than 1 month or older than 15 years old
* Cardiac disease

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients, age ranging from 1 month to 18 years old, meeting the American European Consensus (AECC) definition of ALI and ARDS will be included regardless of etiology of respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
1. Incidence of Pediatric ALI, ARDS and non-ALI/ARDS in Spain based on the AECC and HELP criteria. | One year

SECONDARY OUTCOMES:
Risk factors and causes of ALI/ARDS | One year
  1. Risk factors and causes of ALI/ARDS
  2. Mortality rates of combined ALI/ARDS, established ARDS, and non-ALI/ARDS acute respiratory failure.
  3. Identification of causes of death in ALI and ARDS.
  4. Prognostic factors associated with survival and/or fatal outcome.
  5. Identification of tertiles of clinical data associated with the highest or lowest mortality.
  6. Development of a scoring system for ALI and ARDS prognosis.
  7. Identification of patterns of extrapulmonary organ failure

CONTACTS AND LOCATIONS:
Overall Officials: Kacmarec and Villar Robert and Jesus, Physicians, Principal Investigator — Spanish Intensive Care
Locations (1):
- Cruces Hospital, Barakaldo, Vizcaya, Spain